CLINICAL TRIAL: NCT07091656
Title: Incidence and Risk Factors of Contrast-associated Acute Kidney Injury in Patients Hospitalised After Contrast-enhanced Computed Tomography in the Emergency Department
Brief Title: Contrast-enhanced Computed Tomography and Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Beaujon Hospital (Other)
Responsible Party: Principal Investigator, Prabakar VAITTINADA AYAR, MD, PhD, Beaujon Hospital
Other Study IDs: urgBjNPC-AKI
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Contrast-associated Acute Kidney Injury
Keywords: Acute kidney injury; contrast media; tomography; ontrast-induced nephropathy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: there is no intervention — NO INTERVENTION

SUMMARY:
Rationale and objectives: Since 1930 it has been accepted that intravenous injection of io-dinated contrast agent as part of contrast-enhanced computed tomography (CE-CT) imaging can induce a contrast-associated acute kidney injury (CA-AKI). For the last 10 years, studies have investigated this iatrogenia. However, those works didn't concern French population and particularly patient hospitalised after emergency department (ED) visit.

This study as-sessed the CA-AKI incidence and factor risks in patients hospitalised after a CE-CT in ED.

This was a retrospective cohort observational study in the ED of the Beaujon University Hospital between October 31st 2019 to January 24th 2022.

Patients over 16 years old who presented to the emergency department and underwent an intravenous contrast-enhanced CT were eligible. To be included, patients were required to have at least two creatinine measurements: one taken within 24 hours before CT and a second measurement taken between 48 hours to the seventh day following the initial test. The CT examination had to be performed at Beaujon Hospital with the injection of iodinated contrast agents such as IOMERON® (iomeprol) or XENETIX® (iobitridol).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 16 years old who presented to the emergency department and underwent an intravenous contrast-enhanced CT were eligible. To be included, patients were required to have at least two creatinine measurements: one taken within 24 hours before CT and a sec-ond measurement taken between 48 hours to the seventh day following the initial test. The CT examination had to be performed at Beaujon Hospital with the injection of iodinated contrast agents such as IOMERON® (iomeprol) or XENETIX® (iobitridol).

Exclusion Criteria:

* Patients were excluded from the study if they did not have two creatinine measurements meeting the specified criteria. If multiple contrast-enhanced CT examinations were per-formed within a seven-day period for the same patient, only the first examination was in-cluded in the study, while subsequent scans were excluded.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients over 16 years old who presented to the emergency department and underwent an intravenous contrast-enhanced CT were eligible.
Sampling Method: Non-Probability Sample
Enrollment: 1463 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the occurrence of CA-AKI defined as KDIGO (Kidney Disease Improval Global Outcomes) tage 1 or higher within seven days after contrast-enhanced CT. | BETWEEN 2 and 7 DAYS ATER CT -SCAN

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Beaujon, Clichy, Île-de-France (Paris), France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lecomte E, Vaittinada Ayar P, Vilgrain V, Vaittinada Ayar P. Incidence and risk factors of contrast-associated acute kidney injury in patients hospitalised after contrast-enhanced computed tomography in the emergency department. Int J Emerg Med. 2025 Dec 29;18(1):265. doi: 10.1186/s12245-025-01058-0. PMID 41462065